CLINICAL TRIAL: NCT01894750
Title: Building Skill in Heart Failure Self-Care: A Community Based Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R10-02126; 10CRP4140049 (Other: American Heart Association)
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Self-Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- skill bulding Intevention (Experimental): group-based skill building self-care program
  Interventions: Behavioral: group-based skill building self-care program
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: group-based skill building self-care program
  Arms: skill bulding Intevention

SUMMARY:
The purpose of this study is to pilot and feasibility test an innovative cognitive behavioral intervention to improve heart failure self-care among community dwelling older adults.The primary aim of this study is to test the effect of the intervention on improving heart failure self-care, knowledge and Health related quality of life at 1 month and 3 months. We will test three hypotheses comparing 60 older adults with heart failure randomly assigned to either the intervention or a control group:

Hypothesis 1. Participants in the intervention group will have significantly improved heart failure self-care than control participants.

Hypothesis 2. Participants in the intervention group will have significantly improved knowledge about heart failure and heart failure self-care than control participants.

Hypothesis 3. Participants in the intervention group will have significantly better Health Related Quality of Life than control participants.

A secondary exploratory aim is to assess and describe implementation feasibility of providing a heart failure self-care intervention in a community group setting.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic HF
* able to read and speak English or Spanish
* over age 50

Exclusion Criteria:

* history of prior neurological event (e.g., stroke, head injury, encephalopathy) that could cause dementia
* unable to perform tests or participate in the intervention session (e.g., inability to communicate verbally, major visual impairment, or severe and uncorrected hearing loss).
* living in a nursing home or other long term care facility

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in baseline heart failure self-care score at one month | Change from baseline heart failure self-care at 1 month
  Heart failure self-care is measured by the valid and reliable instrument the Self-Care of Heart Failure Index. Change in scores from baseline at one month will be assessed.
Change in baseline heart failure self-care score at 3 months | Change from baseline heart failure self-care at 3 months
  Heart failure self-care is measured by the valid and reliable instrument the Self-Care of Heart Failure Index. Change in scores from baseline to 3 months will be assessed.

SECONDARY OUTCOMES:
Change in baseline Heart failure knowledge score at 1 month | Change in baseline Heart failure knowledge score at 1 month
  Heart failure knowledge will be measured using the valid and reliable Dutch Heart Failure Knowledge survey. Changes in total score from baseline at 1 month will be assessed.
Change in baseline Heart failure knowledge score at 3 month | Change in baseline Heart failure knowledge score at 3 month
  Heart failure knowledge will be measured using the valid and reliable Dutch Heart Failure Knowledge survey. Changes in total heart failure knowledge score from baseline to 3 months will be assessed.

OTHER OUTCOMES:
Changes in baseline Health related quality of life at 1 month | Changes in baseline health related quality of life at 1 month
  Health related quality of life will be measured using valid and reliable Kansas City Cardiomyopathy Questionnaire. Changes in scores will be assessed from baseline to 3 months
Changes in baseline Health related quality of life at 3 month | Changes in baseline health related quality of life at 3 month
  Health related quality of life will be measured using valid and reliable Kansas City Cardiomyopathy Questionnaire. Changes in scores will be assessed from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Vaughan Dickson, PhD, RN, FAHA, Principal Investigator — NYU College of Nursing
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - NYU Langone Medical Center, New York, New York